CLINICAL TRIAL: NCT00459667
Title: International, Multicenter, Phase IIIb Study of Subcutaneous Every-other-day Treatment of Patients With Relapsing Multiple Sclerosis With (Phase A): Double-blind Betaseron/Betaferon 250µg or 500µg or Open-label Betaseron/Betaferon 250µg and (Phase B): Open-label Betaseron/Betaferon 500µg
Brief Title: BEYOND Follow-up: Betaferon®/Betaseron® Efficacy Yielding Outcomes of a New Dose
Acronym: Beyond
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91656; 2006-005270-47 (EudraCT Number); 309363 (Other: Company internal)
Record Dates: First submitted 2007-04-11; First posted 2007-04-12 (Estimated); Results first posted 2009-08-17 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing multiple sclerosis; interferon beta 1b; Betaferon; Betaseron
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Interferon beta-1b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IFNB-1b 500 mcg (Experimental): Interferon beta 1b ([IFNB 1b] Betaseron) 500 mcg administered s.c. every other day (double blind)
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)
- IFNB-1b 250 mcg (Experimental): Interferon beta 1b ([IFNB 1b] Betaseron) 250 mcg administered s.c. every other day (double blind)
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)
- IFNB-1b 250 mcg* (Experimental): Interferon beta 1b ([IFNB 1b] Betaseron) 250 mcg administered s.c. every other day
  *(Subjects who were administered Copaxone and subjects who had prematurely discontinued medication during BEYOND study.)
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Phase A: 250ug administrated s.c. every other day (double blind). For patients previously randomized in Bayer study 91162 to the same treatment. Phase B: All patients will receive 500µg s.c.every other day (open-label).
  Arms: IFNB-1b 250 mcg
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Phase A: 500ug administrated s.c. every other day (double blind). For patients previously randomized in Bayer study 91162 to the same treatment. Phase B: All patients will receive 500µg s.c.every other day (open-label).
  Arms: IFNB-1b 500 mcg
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Phase A: 250ug administrated s.c. every other day (open-label). For patients previously randomized in Bayer study 91162 to 20mg Copaxone® administrated s.c. once daily and patients with premature discontinuation of study medication during the study 91162.
  Phase B: All patients will receive 500µg s.c.every other day (open-label).
  Arms: IFNB-1b 250 mcg*

SUMMARY:
The BEYOND Follow-Up study will give patients who participated in the preceding BEYOND study the opportunity to continue treatment with the 500µg dose of interferon beta (IFNB) 1b and will further investigate the safety and tolerability profile of interferon beta 1b 500µg during longer-term treatment.

DETAILED DESCRIPTION:
Phase A (3 arm parallel group): All patients randomized during the BEYOND study (Bayer 306440) to either IFNB 1b group (250µg or 500µg) will continue their previously assigned study medication, applying the same level of blinding as during the BEYOND study, All patients randomized during the BEYOND study to Copaxone and all patients with premature discontinuation of study medication during the BEYOND study will receive open-label IFNB 1b 250µg.

Phase B (single arm): All patients will receive open-label IFNB 1b 500µg)

Randomization: No randomization in this trial, patient's allocation in this follow-up study depends only on prior trial groups. The preceding study was randomized.

The trial is sponsored by Bayer Schering Pharma AG, Germany, Bayer HealthCare and Bayer HealthCare Pharmaceuticals Inc.

Secondary outcome measure "Assessment of patient-reported outcomes (FAMS and EQ 5D: The variables FAMS and EQ-5D were not analyzed due to the termination of the study before start of Phase B.

ELIGIBILITY:
Inclusion Criteria:

* Completion of the BEYOND study 306440 as scheduled
* Relapsing multiple sclerosis
* Medical assessment by the investigator that there is no objection to the patient's participation in this trial considering the medical experience from study 306440. Special attention should be given to laboratory abnormalities and clinically relevant liver, renal and bone-marrow dysfunction.
* Females of child-bearing potential:

  * Agreement to practice adequate contraception methods and
  * Negative pregnancy test and
  * No lactation
* Written informed consent

Exclusion Criteria:

* Serious or acute heart diseases
* History of severe depression or suicide attempt
* Epilepsy not adequately controlled by treatment
* Known allergy to IFNs, to human albumin or to mannitol
* Medical, psychiatric or other conditions that compromise the patient's ability to understand the patient information, to give informed consent, to comply with the trial protocol, or to complete the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1420 (Actual)
Dates: Start 2007-05; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (166):
- United States (50):
  - Birmingham, Alabama
  - Cullman, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Berkeley, California
  - La Jolla, California
  - Sacramento, California
  - San Francisco, California
  - Fort Collins, Colorado
  - Newark, Delaware
  - Washington D.C., District of Columbia
  - Maitland, Florida
  - Miami, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - Indianapolis, Indiana
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Shreveport, Louisiana
  - Detroit, Michigan
  - Duluth, Minnesota
  - St Louis, Missouri
  - Henderson, Nevada
  - Reno, Nevada
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Mineola, New York
  - Rochester, New York
  - Stony Brook, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Tualatin, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Fairfax, Virginia
  - Seattle, Washington
  - Tacoma, Washington
  - Milwaukee, Wisconsin
- Argentina (4):
  - Buenos Aires, Buenos Aires
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Córdoba, Córdoba Province
  - Rosario, Santa Fe Province
- Australia (6):
  - Kogarah, New South Wales
  - Fitzroy, Victoria
  - Parkville, Victoria
  - Nedlands, Western Australia
  - Liverpool
  - Wyoming
- Austria (4):
  - Sankt Pölten, Lower Austria
  - Graz
  - Innsbruck
  - Linz
- Belgium (3):
  - Brussels
  - Leuven
  - Melsbroek
- Brazil (6):
  - Curitiba, Paraná
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Campinas, São Paulo
  - São Paulo, São Paulo
- Canada (11):
  - Calgary, Alberta
  - Vancouver, British Columbia
  - Halifax, Nova Scotia
  - London, Ontario
  - Mississauga, Ontario
  - Nepean, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Hull, Quebec
  - Montreal, Quebec
- Aarhus, Denmark
- Finland (2):
  - Oulu
  - Tampere
- France (10):
  - Rennes, Brittany Region
  - Bordeaux, Gironde
  - Clermont-Ferrand
  - Dijon
  - Lille
  - Nancy
  - Nantes
  - Nice
  - Nîmes
  - Toulouse
- Germany (18):
  - Heidelberg, Baden-Wurttemberg
  - Bayreuth, Bavaria
  - Regensburg, Bavaria
  - Hennigsdorf, Brandenburg
  - Hamburg, Hamburg
  - Giessen, Hesse
  - Marburg, Hesse
  - Offenbach, Hesse
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Düsseldorf, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Berlin, State of Berlin
- Greece (2):
  - Athens, Attica
  - Thessaloniki
- Hungary (5):
  - Budapest
  - Győr
  - Miskolc
  - Pécs
  - Zalaegerszeg-Pozva
- Ireland (3):
  - Dublin, Dublin
  - Cork
  - Dublin
- Israel (6):
  - Tel Aviv, Israel
  - Tel Litwinsky, Israel
  - Ẕerifin, Israel
  - Ashkelon
  - Haifa
  - Jerusalem
- Italy (6):
  - Orbassano, Torino
  - Bari
  - Florence
  - Milan
  - Padua
  - Roma
- Riga, Latvia
- Netherlands (3):
  - Breda
  - Nijmegen
  - Sittard
- Bergen, Norway
- Poland (6):
  - Gdansk
  - Katowice
  - Lodz
  - Poznan
  - Warsaw
  - Wroclaw
- Russia (5):
  - Moskva
  - Nizhy Novgorod
  - Novosibirsk
  - Saint Petersburg
  - Yaroslavl
- Slovenia (2):
  - Ljubljana
  - Maribor
- Spain (3):
  - L'Hospitalet de Llobregat, Barcelona
  - Málaga
  - Seville
- Sweden (2):
  - Stockholm
  - Uppsala
- Switzerland (2):
  - Bern
  - Sankt Gallen
- Ukraine (4):
  - Donetsk
  - Kharkiv
  - Kiev
  - Lviv

REFERENCES:
- [Derived] Goodin DS, Hartung HP, O'Connor P, Filippi M, Arnason B, Comi G, Cook S, Jeffery D, Kappos L, Bogumil T, Knappertz V, Sandbrink R, Beckmann K, White R, Petkau J, Pohl C; BEYOND Study Group. Neutralizing antibodies to interferon beta-1b multiple sclerosis: a clinico-radiographic paradox in the BEYOND trial. Mult Scler. 2012 Feb;18(2):181-95. doi: 10.1177/1352458511418629. Epub 2011 Sep 27. PMID 21952094

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible patients for this study included only those who completed the preceding BEYOND study. Patients were enrolled at the conclusion of the preceding study from 03 May 2007 until 14 March 2008. Patients who interrupted study medication in accordance with the investigator were eligible, provided it did not result in premature End of Study.
Pre-assignment Details: All enrolled patients who had been randomized during the predecessor study to IFNB 1b (Interferon 1b) continued on previously double-blinded medication in the BEYOND-FU study; all patients who had been previously randomized to Copaxone and all patients with premature end of study medication received open-label IFNB 1b 250 µg (IFNB 1b 250 µg*).
Period: Overall Study
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg*
Started | 592 | 647 | 181
Study Medication Dispensed | 586 | 645 | 180
Started Treatment | 586 | 644 | 180
Completed | 554 | 600 | 161
Not Completed | 38 | 47 | 20
Not completed — Adverse Event | 9 | 12 | 8
Not completed — Lost to Follow-up | 5 | 9 | 3
Not completed — Pregnancy | 1 | 1 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 5 | 5
Not completed — Other disease modifying treatment | 1 | 2 | 1
Not completed — Other reason (incl. 2 missing subjects) | 12 | 15 | 1
Not completed — No treatment administered | 6 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg* | Total
Number analyzed (Participants) | 586 | 645 | 180 | 1411
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean±Standard Deviation | 36.2 (9.36) | 35.8 (9.17) | 34.9 (9.5) | 35.9 (9.29)
Age, Customized [Number; unit: participants]
  <=18 years | 6 | 5 | 2 | 13
  >18 and <55 years | 580 | 640 | 178 | 1398
  >=55 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 414 | 445 | 113 | 972
  Male | 172 | 200 | 67 | 439

OUTCOME MEASURES:

1. Primary Outcome: Flu-like-syndrome
Description: The variable "Flu-like-syndrome" will consist of a combination of MedDRA terms (Preferred Terms and Lower Level Terms) indicative for this condition.
Time Frame: 309 days
Population: The analysis set used for safety analysis (SAF) comprised 1411 patients. AEs were defined as events with an onset date after the first application of study drug. The incidence rate of Flu-Like-Syndrome with 95% confidence intervals were provided.
Measure: Number; unit: Percentage of participants
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg*
Number analyzed (Participants) | 586 | 645 | 180
Percentage of participants | 17.4 | 15.8 | 31.1
Statistical Analysis 1: Comparison: IFNB-1b 500 mcg; The 95% Confidence Interval was calculated for number of patients w/ Flu-Like-Syndrome; Test type: Superiority or Other; Number of patients w/ Flu-Like-Syndrome = 17.4, 95% CI [14.4 to 20.7]
Statistical Analysis 2: Comparison: IFNB-1b 250 mcg; The 95% Confidence Interval was calculated for number of patients w/ Flu-Like-Syndrome; Test type: Superiority or Other; Number of patients w/ Flu-Like-Syndrome = 15.8, 95% CI [13.1 to 18.9]
Statistical Analysis 3: Comparison: IFNB-1b 250 mcg*; The 95% Confidence Interval was calculated for number of patients w/ Flu-Like-Syndrome; Test type: Superiority or Other; Number of patients w/ Flu-Like-Syndrome = 31.1, 95% CI [24.4 to 38.4]

2. Primary Outcome: Injection-site Reactions
Description: The variable "Injection-site reactions" will consist of a combination of MedDRA terms (Preferred Terms only) indicative for this condition.
Time Frame: 309 days
Population: The analysis set used for safety analysis (SAF) comprised 1411 patients. AEs were defined as events with an onset date after the first application of study drug. The incidence rate of Injection-site reactions with 95% confidence intervals were provided.
Measure: Number; unit: Percentage of participants
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg*
Number analyzed (Participants) | 586 | 645 | 180
Percentage of participants | 31.7 | 26.2 | 31.7
Statistical Analysis 1: Comparison: IFNB-1b 500 mcg; The 95% Confidence Interval was calculated for number of patients w/ Injection-site (IS) reactions; Test type: Superiority or Other; number of patients w/ IS reactions. = 31.7, 95% CI [28.0 to 35.7]
Statistical Analysis 2: Comparison: IFNB-1b 250 mcg; The 95% Confidence Interval was calculated for number of patients w/ Injection-site (IS) reactions; Test type: Superiority or Other; number of patients w/ IS reactions. = 26.2, 95% CI [22.8 to 29.8]
Statistical Analysis 3: Comparison: IFNB-1b 250 mcg*; The 95% Confidence Interval was calculated for number of patients w/ Injection-site (IS) reactions; Test type: Superiority or Other; number of patients w/ IS reactions. = 31.7, 95% CI [24.9 to 39.0]

3. Primary Outcome: Liver Enzyme Elevations
Description: The variable "Liver enzyme elevations" will consist of a combination of MedDRA terms (Preferred Terms only) indicative for this condition.
Time Frame: 309 days
Population: The analysis set used for safety analysis (SAF) comprised 1411 patients. AEs were defined as events with an onset date after the first application of study drug. The incidence rate of liver enzyme elevations were provided.
Measure: Number; unit: Percentage of participants
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg*
Number analyzed (Participants) | 586 | 645 | 180
Percentage of participants
  GGT increased | 2.7 | 1.2 | 3.9
  AST increased | 2.0 | 1.4 | 3.9
  ALT increased | 2.6 | 1.7 | 4.4

4. Primary Outcome: Hematological Abnormalities
Description: The variable "Hematological abnormalities" will consist of a combination of MedDRA terms (Preferred Terms only) indicative for this condition.
Time Frame: 309 days
Population: The analysis set used for safety analysis (SAF) comprised 1411 patients. AEs were defined as events with an onset date after the first application of study drug. The incidence rate of hematological abnormalities were provided.
Measure: Number; unit: Percentage of participants
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg*
Number analyzed (Participants) | 586 | 645 | 180
Percentage of participants
  White blood cells decreased | 0.5 | 1.9 | 1.7
  Neutrophil count decreased | 0.5 | 1.2 | 2.2
  Lymphocyte count decreased | 1.5 | 0.6 | 0
  Platelet count decreased | 0.7 | 0.2 | 0.6
  Hemoglobin decreased | 1.2 | 1.1 | 0

5. Secondary Outcome: Percentage of Patients With Neutralizing Antibody Titer to IFNB-1b of Different Cut-off Values
Description: Serum samples of about 8 mL for analysis of neutralizing antibodies (NAbs) to interferon (IFN) beta-1b were drawn at Baseline, Week 26 and the EOS visit.
Time Frame: 309 days
Population: For the NAb analyses data were provided for 572 patients at Baseline, 238 at Week 26 and 1261 at EOS. The patients missing to the total number of 1411 patients had no data at the respective visits (table shows number of patients with positive titer in the extension treatment cohorts; the analyses provide frequencies of positive titers).
Measure: Number; unit: Percentage of participants
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg*
Number analyzed (Participants) | 527 | 571 | 163
Percentage of participants
  NAbs titer, cut-off value 20 NU/ml | 26.6 | 21.7 | 16.6
  NAbs titer, cut-off value 100 NU/ml | 16.5 | 12.4 | 2.5
  NAbs titer, cut-off value 400 NU/ml | 10.8 | 6.1 | 0

ADVERSE EVENTS:
Arm/Group | IFNB-1b 500 mcg | IFNB-1b 250 mcg | IFNB-1b 250 mcg*
Serious Adverse Events (participants affected / at risk) | 11/586 | 16/645 | 6/180
Other Adverse Events (participants affected / at risk) | 455/586 | 467/645 | 136/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IFNB-1b 500 mcg (N=586) | IFNB-1b 250 mcg (N=645) | IFNB-1b 250 mcg* (N=180)
Carotid artery stenosis (Nervous system disorders) | 0 | 1 | 0
Multiple Sclerosis (Nervous system disorders) | 1 | 0 | 0
Optic neuritis (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0
Bladder catheter replacement (Surgical and medical procedures) | 0 | 0 | 1
Elective surgery (Surgical and medical procedures) | 1 | 0 | 2
Rehabilitation therapy (Surgical and medical procedures) | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Dandy-Walker syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Papillitis (General disorders) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Injection site cellulitis (Infections and infestations) | 0 | 1 | 0
Arteriogram coronary (Investigations) | 0 | 1 | 0
Platelet aggregation (Investigations) | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intra-uterine death (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Renal failure actue (Renal and urinary disorders) | 0 | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IFNB-1b 500 mcg (N=586) | IFNB-1b 250 mcg (N=645) | IFNB-1b 250 mcg* (N=180)
Astenia (General disorders) | 10 | 14 | 0
Chills (General disorders) | 4 | 7 | 4
Fatigue (General disorders) | 89 | 89 | 23
Influenza like illness (General disorders) | 72 | 62 | 37
Injection site bruising (General disorders) | 18 | 12 | 3
Injection site erythema (General disorders) | 70 | 73 | 17
Injection site induration (General disorders) | 3 | 2 | 4
Injection site mass (General disorders) | 4 | 1 | 4
Injection site nodule (General disorders) | 0 | 1 | 5
Injection site pain (General disorders) | 25 | 17 | 11
Injection site reaction (General disorders) | 80 | 70 | 20
Pain (General disorders) | 15 | 6 | 3
Pyrexia (General disorders) | 6 | 2 | 10
Dizziness (Nervous system disorders) | 16 | 13 | 3
Headache (Nervous system disorders) | 72 | 89 | 26
Hypoaesthesia (Nervous system disorders) | 19 | 23 | 7
Migraine (Nervous system disorders) | 8 | 15 | 2
Multiple sclerosis relapse (Nervous system disorders) | 45 | 71 | 13
Muscle spasticity (Nervous system disorders) | 11 | 11 | 7
Paraesthesia (Nervous system disorders) | 26 | 43 | 12
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 33 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 35 | 30 | 6
Muscle spams (Musculoskeletal and connective tissue disorders) | 26 | 23 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 | 14 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 13 | 19 | 7
Pain in extremitiy (Musculoskeletal and connective tissue disorders) | 28 | 29 | 14
Nasopharyngitis (Infections and infestations) | 11 | 21 | 8
Sinusitis (Infections and infestations) | 5 | 8 | 4
Upper respiratory tract infection (Infections and infestations) | 6 | 12 | 10
Urinary tract infection (Infections and infestations) | 9 | 9 | 8
Alanine aminotransferase increased (Investigations) | 15 | 11 | 8
Aspartate aminotransferase increased (Investigations) | 12 | 9 | 7
Gamma-glutamyltransferase increased (Investigations) | 16 | 8 | 7
Neutrophil count decreased (Investigations) | 3 | 8 | 4
Anxiety (Psychiatric disorders) | 25 | 27 | 6
Depression (Psychiatric disorders) | 56 | 60 | 23
Constipation (Gastrointestinal disorders) | 11 | 12 | 7
Micturition urgency (Renal and urinary disorders) | 13 | 6 | 2
Leukopenia (Blood and lymphatic system disorders) | 15 | 17 | 5
Neutropenia (Blood and lymphatic system disorders) | 14 | 5 | 3
Hypertension (Vascular disorders) | 22 | 26 | 7
Vision blurred (Eye disorders) | 9 | 12 | 4
Vertigo (Ear and labyrinth disorders) | 11 | 9 | 4
Nausea (Gastrointestinal disorders) | 7 | 9 | 6
Injection site atrophy (General disorders) | 0 | 1 | 4
Oedema peripheral (General disorders) | 2 | 3 | 4
Pharyngitis (Infections and infestations) | 4 | 2 | 4
Burning sensation (Nervous system disorders) | 2 | 8 | 5
Urinary incontinence (Renal and urinary disorders) | 4 | 7 | 4
Menopausal symptoms (Reproductive system and breast disorders) | 3 | 1 | 4
Insomnia (Psychiatric disorders) | 23 | 35 | 7

LIMITATIONS AND CAVEATS:
Due to the termination of the study before start of Phase B according to protocol defined stopping rules, functional assessments of multiple sclerosis (FAMS) and EuroQoL (EQ-5D) were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor is interested in the publication of the results of every study it performs. As some of the information concerning the study drug and the sponsor's development activities may be strictly confidential, any publication manuscript (including conference contributions, etc.) must first be reviewed by the sponsor before its submission or presentation. Publication of subgroup data and single center data shall not be performed until the complete study has been published.